CLINICAL TRIAL: NCT06851143
Title: 18F-DPA-714 PET/MR in Dysfunctional Brain Diseases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20252023
Record Dates: First submitted 2025-02-19; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Brain Disease
Keywords: 18F-DPA-714 PET/MR; cognitive impairment; dyskinesia; Disorders of consciousness; Autoimmune encephalitis
MeSH Terms: conditions — Brain Diseases; Cognitive Dysfunction; Dyskinesias; Consciousness Disorders; Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Comparative study of different groups (Other): This study is planned to include approximately 25 normal volunteers and 40 patients with dysfunctional brain diseases. The screened subjects will undergo multimodal imaging data acquisition using integrated PET/MR (GE Signa). The SUV ratio (SUVR) of each brain region will be obtained using the cerebellum as a reference, and differences in [18F]DPA-714 uptake between patients and normal controls will be compared using voxel-based imaging analysis. PCA-based analysis of the distribution pattern of TSPO radioabnormalities in different types of patients. Pearson correlation-based analysis of the correlation between neuroimmune activation and structural and functional parameters.
  Interventions: Diagnostic Test: 18F-DPA-714 PET/MR scan

INTERVENTIONS:
Diagnostic Test: 18F-DPA-714 PET/MR scan — Saline intravenous solution of 18F-DPA-714 administered at 0.1 mCi/kg by bodyweight

SUMMARY:
This is a diagnostic pilot study that recruited 25 normal volunteers and 40 patients with dysfunctional brain diseases and performed 18F-DPA-714 PET/MR imaging to evaluate the correlation between the multimodal imaging features of dysfunctional brain diseases, to explore the potential pathological mechanisms of neuroimmune activation, and to further analyse the value of PET/MR-based multimodal imaging in the diagnosis and differential diagnosis of dysfunctional brain diseases. and further analyse the diagnostic and differential diagnostic value of PET/MR-based multimodal imaging in dysfunctional brain diseases.

ELIGIBILITY:
Inclusion Criteria:

* Dysfunctional disorders diagnosed according to the guidelines include: cognitive disorders, movement disorders, disorders of consciousness-like disorders, and autoimmune encephalitis. Signing the PET/MR informed consent form to volunteer for this study

Exclusion Criteria:

* Minors, pregnant women, nursing mothers, those with severe liver or kidney insufficiency, history of allergy to contrast media or other drugs. Diagnosis of viral encephalitis, acute myelitis, idiopathic epilepsy, antibody-negative AIE; diagnosis of any major disease; history of alcohol or drug abuse/dependence; history of cardiorespiratory disease, oncology, haematological disorders, poorly controlled chronic diseases; contraindications to PET/MR examination. History of head trauma, history of surgery. History of other neurological disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Standardized uptake value (SUVmax) | 1 day from injection of the tracer

IPD SHARING:
Plan to Share IPD: No